CLINICAL TRIAL: NCT02317536
Title: A Randomized Double-Blind, Placebo-Controlled Pilot Clinical Trial to Evaluate the Relative Efficacy of Two Carnitine-Based Products Purported to Promote Muscle Anabolism in Healthy Older Adults
Brief Title: A Pilot Clinical Trial on the Efficacy of Two Carnitine-Based Products on Muscle Function in Healthy Older Adults
Acronym: 15CAHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Lonza Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 15CAHL
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Muscle Function
Keywords: Muscle function; L-Carnitine; Carnipure; DXA; anabolism; 6 minute walk; dynamometry; muscle biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carnipure Product 1 (Experimental): Carnitine-based product 1, subjects will take one dose once daily for 56 days.
  Interventions: Dietary Supplement: Carnipure Product 1
- Carnipure Product 2 (Experimental): Carnitine-based product 2, subjects will take one dose once daily for 56 days.
  Interventions: Dietary Supplement: Carnipure Product 2
- Placebo (Placebo Comparator): Placebo, subjects will take one dose once daily for 56 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Carnipure Product 1
  Arms: Carnipure Product 1
Dietary Supplement: Carnipure Product 2
  Arms: Carnipure Product 2
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study evaluates two L-Carnitine-based products on muscle function in healthy older adults (55 to 70 years old). These products are suspected to improve muscle function and possibly promote building of muscle mass. One third of the subjects will be on Carnipure Product 1, one third will be on Carnipure Product 2 and one third will be on placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, aged 55 to 70 years
* BMI of 21 kg/m2 to 33 kg/m2
* Subjects in good physical condition such that they can perform exercise testing safely, as determined by the Qualified Investigator based on medical history, physical examination, electrocardiogram and laboratory results
* Subjects who are sedentary and not currently engaging in any regular exercise.
* Subjects who agree to maintain their current level of activity and current dietary habits throughout the trial period.
* Subjects who have given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Subjects who are smokers or have been a smoker within the past 1 year from screening.
* Subjects who are pregnant or breastfeeding
* Subjects who have experienced weight loss or gain of greater than 4.5 kg (approximately 10 lbs) within 3 months of randomization
* Subjects diagnosed with active heart disease
* Subjects with uncontrolled hypertension (≥ 140 mmHg)
* Subjects with renal or hepatic impairment or disease
* Subjects with any major diseases of the gastrointestinal, pulmonary or endocrine systems
* Subjects with a history of seizures
* Subjects with Type I or Type II Diabetes
* Subjects with active cancer (excluding basal cell carcinoma)
* Subjects with neurological or significant psychiatric illnesses, including Parkinson's disease and bi-polar disorder
* Subjects with unstable thyroid disease
* Subjects who are immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis)
* Subjects with metal fixation plates or screws from a previous surgery
* Subjects who are taking oral anticoagulants (blood thinners) such as warfarin (Coumadin) or Dabigatran (Pradaxa) or antiplatelet agents such as Clopidogrel (Plavix)
* Subjects who are regularly taking NSAID medications such as aspirin, must stop at least one week prior to the micro-needle muscle biopsy procedures.
* Subjects with a known allergy to anesthetic
* Subjects who currently experience any medical condition that interferes with the ability to undergo physical strength testing during the study
* Subjects currently taking NHPs must have been using their current dosing regimen for at least one month prior to baseline and must maintain their current dosing regimen throughout the trial and must not begin taking any new NHPs throughout the trial. If the subject wishes to stop taking the NHP prior to beginning the trial, they must do so at least 1 week prior to randomization.
* Subjects who use illicit drugs or have a history of alcohol or drug abuse within the past 6 months
* Subjects who currently consume greater than 2 standard alcoholic drinks per day.
* Subjects who have participated in a clinical research trial within 30 days prior to randomization.
* Subjects with an allergy or sensitivity to the investigational product ingredient.
* Subjects who are cognitively impaired and/or who are unable to give informed consent
* Subjects who have abnormal laboratory results or any other medical or psychological condition which, in the opinion of the Qualified Investigator, may adversely affect the subjects ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percent Change in Muscle Function Composite Endpoint from Baseline to Day 57 of subjects administer Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  A composite endpoint determined by multiplying the values of Lean Body Mass (as assessed by DXA, kg), and functional muscle strength (as assessed by 6 Minute Walk Test, metres; Lower Body Dynamometry, kg; Upper Body Dynamometry, kg). Percent change from baseline to day 57 will be derived.

SECONDARY OUTCOMES:
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  Functional lower body strength will be determined using a hand-held dynamometer to measure leg extension resistance (kg of resistance).
Changes in functional upper body strength from baseline to Day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  Functional upper body strength will be determined using a grip strength dynamometer to measure grip strength resistance (kg of resistance).
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  Functional lower body strength will be assessed using the 6 Minute Walk Test to determine the distance walked over 6 minutes (metres).
Changes in Quality of Life questionnaire score from baseline to day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  Assessed using the RAND SF-36 questionnaire
Changes in Lean Body Mass from baseline to day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Baseline and Day 57
  Lean Body Mass measured by DXA scan

OTHER OUTCOMES:
Changes in muscle metabolism from baseline to day 57 in subjects administered Carnipure Product 2 versus Placebo | Baseline and Day 57
  Assessed by laboratory analysis of muscle biopsy samples collected at baseline (pre-strength testing) and Day 57 (pre and post-strength testing)
Percent Change in Muscle Function Composite Endpoint from Baseline to Day 57 of subjects administer Carnipure Product 1 versus those administered Placebo | Baseline and Day 57
  A composite endpoint determined by multiplying the values of Lean Body Mass (as assessed by DXA, kg), and functional muscle strength (as assessed by 6 Minute Walk Test, metres; Lower Body Dynamometry, kg; Upper Body Dynamometry, kg). Percent change from baseline to day 57 will be derived.
Percent Change in Muscle Function Composite Endpoint from Baseline to Day 57 of subjects administer Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  A composite endpoint determined by multiplying the values of Lean Body Mass (as assessed by DXA, kg), and functional muscle strength (as assessed by 6 Minute Walk Test, metres; Lower Body Dynamometry, kg; Upper Body Dynamometry, kg). Percent change from baseline to day 57 will be derived.
Changes in Lean Body Mass from baseline to day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Baseline and Day 57
  Lean Body Mass measured by DXA scan
Changes in Lean Body Mass from baseline to day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  Lean Body Mass measured by DXA scan
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Baseline to Day 57
  Functional lower body strength will be determined using a hand-held dynamometer to measure leg extension resistance (kg of resistance).
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  Functional lower body strength will be determined using a hand-held dynamometer to measure leg extension resistance (kg of resistance).
Changes in functional upper body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Baseline and Day 57
  Functional upper body strength will be determined using a grip strength dynamometer to measure grip strength resistance (kg of resistance).
Changes in functional upper body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  Functional upper body strength will be determined using a grip strength dynamometer to measure grip strength resistance (kg of resistance).
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Baseline and Day 57
  Functional lower body strength will be assessed using the 6 Minute Walk Test to determine the distance walked over 6 minutes (metres).
Changes in functional lower body strength from baseline to Day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  Functional lower body strength will be assessed using the 6 Minute Walk Test to determine the distance walked over 6 minutes (metres).
Changes in Quality of Life questionnaire score from baseline to day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Baseline and Day 57
  Assessed using the RAND SF-36 questionnaire
Changes in Quality of Life questionnaire score from baseline to day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Baseline and Day 57
  Assessed using the RAND SF-36 questionnaire
Changes in muscle metabolism from baseline to day 57 in subjects administered Carnipure Product 1 versus Placebo | Baseline and Day 57
  Assessed by laboratory analysis of muscle biopsy samples collected at baseline (pre-strength testing) and Day 57 (pre and post-strength testing)
Changes in muscle metabolism from baseline to day 57 in subjects administered Carnipure Product 1 versus Carnipure Product 2 | Baseline and Day 57
  Assessed by laboratory analysis of muscle biopsy samples collected at baseline (pre-strength testing) and Day 57 (pre and post-strength testing)
Changes in vital signs from baseline to day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Screening to Day 57
  Blood pressure, heart rate, BMI, electrocardiogram
Changes in vital signs from baseline to day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Screening to Day 57
  Blood pressure, heart rate, BMI, electrocardiogram
Changes in vital signs from screening to day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Screening to Day 57
  Blood pressure, heart rate, BMI, electrocardiogram
Changes in hematology and clinical chemistry from screening to Day 57 in subjects administered Carnipure Product 2 versus those administered Placebo | Screening and Day 57
  CBC, electrolytes, glucose, creatinine, AST, ALT, GGT, bilirubin
Changes in hematology and clinical chemistry from screening to Day 57 in subjects administered Carnipure Product 1 versus those administered Placebo | Screening and Day 57
  CBC, electrolytes, glucose, creatinine, AST, ALT, GGT, bilirubin
Changes in hematology and clinical chemistry from screening to Day 57 in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | Screening and Day 57
  CBC, electrolytes, glucose, creatinine, AST, ALT, GGT, bilirubin
Number of adverse events experienced in subjects administered Carnipure Product 2 versus those administered Placebo | 57 days
Number of adverse events experienced in subjects administered Carnipure Product 1 versus those administered Placebo | 57 days
Number of adverse events experienced in subjects administered Carnipure Product 1 versus those administered Carnipure Product 2 | 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada